CLINICAL TRIAL: NCT05490654
Title: Tailored Abdominal Massage Treatment for Constipation in Adults With Learning Disabilities- A Feasibility Study and Pilot Trial
Brief Title: Abdominal Massage for People With Learning Disabilities and Constipation
Acronym: AMID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: Baily Thomas Charitable Fund (Unknown); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 307439
Record Dates: First submitted 2022-07-26; First posted 2022-08-08 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Single-centre feasibility randomised controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Massage (Experimental): Study participants who will receive abdominal massage by manual or device delivered for 6 weeks
  Interventions: Procedure: Abdominal Massage
- Control (No Intervention): Participants who will have no change to their normal treatment regime

INTERVENTIONS:
Procedure: Abdominal Massage — Abdominal Massage delivered by manual method or by Mowoot device
  Arms: Abdominal Massage

SUMMARY:
Background and study aims:

Constipation, which is difficulty going to the toilet to do a 'poo' is common in adults with learning disabilities (LD), but there is not a lot of knowledge (information) about the best way to help treat constipation experienced by adults with learning disabilities. Adults with learning disabilities who have constipation should be assessed and treated. There is knowledge to suggest that abdominal massage may help some people with constipation so that people with constipation can go to the toilet more easily.

There is also knowledge to suggest that the use of a device to do the massage may be as beneficial as getting a carer to do it for the participant.

This research wants to invite 40 adults with learning disabilities with constipation to take part. 30 will be offered the abdominal massage, either by a carer or the device, and 10 will not be offered the massage. However, the participants will be shown how to do it at the end of the study.

This research wants to find out if people with LD are willing to take part in such a study and if the participants are more willing to let a carer do the massage, or would rather use the device. It is also important that the investigators know if the participants who are in the group not getting the massage are willing to continue in the research. Taking part for 6 weeks will provide the investigators with this important information before the investigators undertake a much larger study which the investigators need to do to find out if it helps with constipation.

ELIGIBILITY:
Inclusion Criteria:

1. A person with a Learning Disability who is known to suffer from constipation including:

1a-those on long term laxatives but still prone to constipation

1b- those who have been admitted to hospital due to impaction

1c- those who use enemas regularly but still have emptying problems.

Exclusion Criteria:

1. A history of malignant bowel obstructions or abdominal growth
2. A history of inflammatory bowel disease of the intestine e.g. Chron's disease
3. Unstable spinal surgery
4. Recent scarring or abdominal surgery
5. Abdominal skin lesions
6. Abdominal hernia
7. Pregnancy
8. Indwelling catheter
9. Increased sensitivity to touch
10. Has undertaken Abdominal Massage within the last 3 months.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Feasibility of the abdominal massage intervention | 6 weeks
  Feasibility Questionnaire (Non- validated) to determine the acceptability of the intervention. Content analysis of free text and scoring of 0-5 Likert scale for level of confidence for posed questions with 5 being highly confident and 0 having no confidence.

SECONDARY OUTCOMES:
Knowles-Eccersley-Scott Symptom Score (KESS) | 6 weeks
  The Knowles-Eccersley-Scott Symptom Score will assess degree and impact of constipation and be completed before and after the intervention. 11 scored questions with score values of Minimum 1 and maximum of 5. The higher score indicates the higher degree of severity.
7 Day Bowel Diary (Non-validated scoring tool) | 6 weeks
  7 day Bowel Diary completed before and after the intervention. Scoring indicates the frequency of stools per day for 7 days with the higher number indicating a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Greater Glasgow & Clyde, Glasgow, Strathclyde, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Any request for participant data can be made to Dr Kirsteen Goodman